CLINICAL TRIAL: NCT04942600
Title: Assessing the Behavioural and Electrophysiological Effects of Repetitive Transcranial Magnetic Stimulation on "Intention" vs "Overt Action" in Patients With Functional Neurological Disorders
Brief Title: Behavioural and Electrophysiological Effects of rTMS in Functional Neurological Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: University of Winnipeg (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HS24851 (B2021:033)
Record Dates: First submitted 2021-06-11; First posted 2021-06-28 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Functional Neurological Disorder
MeSH Terms: conditions — Conversion Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Repetitive Transcranial Magnetic Stimulation (rTMS) (Experimental): 1 session (3,000 pulses) of high-frequency (10Hz) repetitive stimulation applied over the right temporal parietal junction (TPJ) gyrus in individuals with Functional Neurological Disorder using a MagStim Rapid2 Transcranial Magnetic Simulation machine.
  Interventions: Device: MagStim Rapid2 Transcranial Magnetic Simulation

INTERVENTIONS:
Device: MagStim Rapid2 Transcranial Magnetic Simulation — A non-invasive method of brain stimulation

SUMMARY:
The purpose of this study is to better understand Functional Neurological Disorders (FND) by measuring movement timing and brain activity in patients with FND during deliberate movements and when expressing an 'intention' to move. This investigation will use non-invasive brain stimulation to investigate the role of the temporal-occipital-parietal junction in FND.

DETAILED DESCRIPTION:
This study seeks to improve our neurophysiological understanding of Functional Neurological Disorders (FND) by measuring movement timing and brain activity while individuals with FND perform a simple pointing task.

Behavioural (timing of arm and finger movement) and electrophysiological (electroencephalography; EEG) measures will be collected both at rest and while participants perform a voluntary movement task designed to discriminate between brain events related to intention vs. overt action.

Furthermore, this study will investigate the ability of a non-invasive brain stimulation technique called repetitive transcranial magnetic stimulation (rTMS) to alter brain activity in the temporal-occipital-parietal junction (TPJ), a region known to be hypo-active in individuals with FND. Tasks and cortical recordings will be repeated following rTMS to determine the effect of brain stimulation on behaviour and brain activity.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Functional Neurological Disorder with motor symptoms.

Exclusion Criteria:

* Presence of another comorbid psychiatric disorder;
* Any contraindication for rTMS (e.g., implanted metal devices; cardiac pacemaker or pacemaker wires; neurostimulators; implanted pumps, metal in the body [rods, plates, screws, shrapnel, dentures, IUD] or metallic particles in the body, surgical clips in the head, previous neurosurgery, cochlear implants, prosthetic heart valves);
* Currently pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Change in relative timing of intention-to-act vs action production | 1 hour: Immediately prior to and following one session of rTMS
  Assessment of change in the lag time between intended and actual action production during pointing and stimulus response tasks.
Change in resting state activity in temporal-parietal junction brain region | 1 hour: Immediately prior to and following one session of rTMS
  Assessment of changes in EEG brain activity readings when participants are at rest at various frequencies, primarily targeting delta/theta bands.

SECONDARY OUTCOMES:
Change in brain activity related to 'intention to act' | 1 hour: Immediately prior to and following one session of rTMS
  Assessment of changes in ERP waveform amplitude related to the 'intention to act' time-stamp during the movement task.
Change in brain activity related to motor production | 1 hour: Immediately prior to and following one session of rTMS
  Assessment of changes in ERP waveform amplitude related to the 'motor production' time-stamp during the movement task.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Bolster, PhD, Principal Investigator — University of Winnipeg; Mandana Modirrousta, MD PhD, Principal Investigator — University of Manitoba
Locations (1):
- St. Boniface Hospital, Winnipeg, Manitoba, Canada